CLINICAL TRIAL: NCT01148680
Title: Randomized Controlled Trial Comparing the Metabolic Efficiency of Allogeneic Pancreatic Islet Transplantation to Intensive Insulin Therapy for the Treatment of Type 1 Diabetes
Brief Title: Trial Comparing Metabolic Efficiency of Islet Graft to Intensive Insulin Therapy for Type 1 Diabetes's Treatment
Acronym: TRIMECO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 08 31
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Islet Cell Transplantation; Metabolic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Metabolic Diseases; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate registration on islet graft list (Experimental): group 1 'immediate registration on infusion waiting list' : patients who will be immediately registrated on islet cell infusion waiting list after randomization.
  Intervention : Procedure/surgery (islet graft)
  Interventions: Biological: Islet Graft
- delayed registration on islet graft list (Active Comparator): group 2 'delayed registration on infusion waiting list' : patients who will be registrated 6 months later on islet cell infusion waiting list after randomization.
  Intervention : Procedure/surgery (islet graft)
  Interventions: Biological: Islet Graft

INTERVENTIONS:
Biological: Islet Graft — Iterative injection of pancreatic islets (minimum: 250,000 IEQ / injection or 3500 IEQ / kg / injection) with a threshold required total of 11,000 IEQ / kg in 2 or 3 injections per patient)
  Other Names: human pancreatic islet transplantation

SUMMARY:
Efficacy of pancreatic islet transplantation at 6 months compared to an intensive insulin therapy for 2 categories of patients: patients with unstable diabetes and patients who underwent kidney transplantation.

DETAILED DESCRIPTION:
Efficacy of pancreatic islet transplantation at 6 months compared to an intensive insulin therapy for 2 categories of patients: patients with unstable type 1 diabetes versus patients with unstable type 1 diabetes and who underwent kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 diabetes or C-peptide negative diabetes Diabetes duration > 5 years
* No residual insulin secretion (plasmatic basal and stimulated C-peptide < 0.3 ng/ml)
* HbA1c considered acceptable by the selection committee
* Insulin needs < 0.85 IU/kg/day
* Islet cell infusion after kidney graft

  * Patient with terminal renal failure and functional kidney graft for at least 6 months (creatinine clearance greater than or equal to 35 ml/min)
  * Patient whose glycaemic control obtained with insulin therapy could threaten kidney graft survival and/or significantly alter quality of life. This situation is assessed by a diabetologist
* Islet cell infusion only: patient with major glycaemic variability despite proper intensive insulin therapy, closely monitored by a diabetologist. Poor glucose control, assessed by a diabetologist, endangers the patient's life and/or significantly alters personal, social, professional and family quality of life. At least one of these criteria must be fulfilled :

  * Hypoglycaemia unawareness, blood glucose level < 3mmol/L or 0.54 mg/L
  * At least 2 severe hypoglycaemia events (defined by the necessity of a third party's assistance) per year or a ketoacidosis requiring patient's hospitalization during the last year.
  * Impairment of quality of life or life-threat for patient or other persons, or progressive complications despite optimal insulin therapy
* Social Security membership or benefit from Social Welfare

Exclusion Criteria:

* Age< 18 and > 65
* Diabetes duration < 5 years
* Criteria specifically related to the islet intraportal injection procedure: hemostasis problem, haemoglobin level < 11g/dL for women and <12g/dL for men, abnormalities of complete blood count, documented liver pathology (alkaline phosphatases, gamma GT, transaminases levels over twice normal values) ; pancreatitis history, gallbladder stones that could potentially migrate; HLA hyperimmunisation (PRA >20%).
* Criteria related to diabetes complications :

  * Non-stabilized proliferating diabetic retinopathy
  * Creatininaemia > 16 mg/dL
* Exclusion criteria non-specifically related to islet infusion: evolutive vascular disease, evolutive cardiopathy (especially myocardial infarction less than 6 months ago, cerebrovascular stroke less than 6 months ago, evolutive arteritis with trophic disorders) ; systemic infection including hepatitis C and HIV ; leuconeutropenia ; thrombocytopenia, non-stabilized neoplastic pathology ; pregnancy or project of pregnancy within the next 24 months ; poor therapeutic compliance
* Criteria related to immunosuppressive protocol : renal failure (glomerular filtration < 35 ml/min/1.73 m²) and/or proteinuria > 0.5 g/24h ; non-treated hyperlipidemia (LDL-C > 130 mg/dL) ; blood pressure > 160/100 mmHg
* Clinical insulin resistance : assessed by patient's weight, BMI and exogenous insulin requirements (BMI > 30 kg/m² or insulin dose > 0.85 UI/kg/day)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
ß score evaluation 6 months after first infusion (group 1 'immediate registration on infusion waiting list') or 6 months after inclusion (group 2: 'delayed registration on infusion waiting list') | 6 months after first infusion (group 1) or 6 months after inclusion (group 2)
  Metabolism evaluated by ß score. This score uses 4 intermediate scores ranging from 0 to 2 associated with the following 4 indicators: HbA1c, basal C peptide (or stimulated C-peptide), daily insulin dose (U/kg) or intake of oral antidiabetic drugs and fasting glycaemia. The total of the intermediate scores ranges from 0 to 8. Islet graft will be considered as successful if the ß score is equal to or greater than 6

SECONDARY OUTCOMES:
Evaluation of metabolism indicators : ß-score and individual analysis of the 4 components of the ß-score | 6 and 12 months
  Metabolism indicators at 6 and 12 months : ß-score (quantitative analysis by mean score comparison), individual analysis of the 4 components of the ß-score (HbA1c, basal C peptide (or stimulated C-peptide), daily insulin dose (U/kg) or intake of oral antidiabetic drugs and fasting glycaemia), lability index, ADRR score, Clarke score
Measure of quality of life (SF36, DQOL, DHP) | at inclusion time, at 6 months and at 12 months after first infusion (group 1) or after inclusion (group 2)
  Measure of quality of life (SF36, DQOL, DHP) for Group 1 ('immediate registration on infusion waiting list'): at inclusion time, at 6 months and at 12 months after first infusion For Group 2 ('delayed registration on infusion waiting list'): at inclusion time, 6 months after inclusion, at 6 months and at 12 months after first infusion
Cost evaluation of islet cell infusion | 6 months
  Cost comparison between islet cell infusion (group 1 'immediate registration on infusion waiting list')and intensive insulin therapy (group 2 'delayed registration on infusion waiting list') at 6 months, from a hospital perspective as well as a health-insurance system perspective
Evaluation of side effects and iatrogenic effects | at 6 months and 12 months after infusion
  Evaluation of side effects and iatrogenic effects at 6 months and 12 months after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, Pr, Principal Investigator — University Hospital, Grenoble
Locations (9):
- France (8):
  - University Hospital, Department of Endocrinology, Strasbourg, Alsace
  - University Hospital, Department of Endocrinology, Grenoble, Auvergne-Rhône-Alpes
  - HCL Sud, Department of Endocrinology, Lyon, Auvergne-Rhône-Alpes
  - University Hospital Gabriel Montpied, Department of Endocrinology, Clermont-Ferrand, Auvergne
  - University Hospital Besançon, Department of Endocrinology, Besançon, Franche-Comté
  - University Hospital, Department of General Surgery and Endocrinology, Lille, Hauts-de-France
  - University Hospital, Department of Endocrinology, Montpellier, Languedoc-Roussillon
  - University Hospital, Department of Endocrinology, Nancy, Lorraine
- Hopitaux Universitaires de Genève, Department of Visceral Surgery and Transplant, Geneva, Switzerland

REFERENCES:
- [Background] Alejandro R, Barton FB, Hering BJ, Wease S; Collaborative Islet Transplant Registry Investigators. 2008 Update from the Collaborative Islet Transplant Registry. Transplantation. 2008 Dec 27;86(12):1783-8. doi: 10.1097/TP.0b013e3181913f6a. PMID 19104422
- [Background] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- [Background] Badet L, Benhamou PY, Wojtusciszyn A, Baertschiger R, Milliat-Guittard L, Kessler L, Penfornis A, Thivolet C, Renard E, Bosco D, Morel P, Morelon E, Bayle F, Colin C, Berney T; GRAGIL Group. Expectations and strategies regarding islet transplantation: metabolic data from the GRAGIL 2 trial. Transplantation. 2007 Jul 15;84(1):89-96. doi: 10.1097/01.tp.0000268511.64428.d8. PMID 17627243
- [Background] Vantyghem MC, Kerr-Conte J, Arnalsteen L, Sergent G, Defrance F, Gmyr V, Declerck N, Raverdy V, Vandewalle B, Pigny P, Noel C, Pattou F. Primary graft function, metabolic control, and graft survival after islet transplantation. Diabetes Care. 2009 Aug;32(8):1473-8. doi: 10.2337/dc08-1685. PMID 19638525
- [Background] Ryan EA, Paty BW, Senior PA, Lakey JR, Bigam D, Shapiro AM. Beta-score: an assessment of beta-cell function after islet transplantation. Diabetes Care. 2005 Feb;28(2):343-7. doi: 10.2337/diacare.28.2.343. PMID 15677790
- [Derived] Bahougne T, Olagne J, Munch M, Braun-Parvez L, Chenard MP, Fremeaux-Bacchi V, Caillard S, Baltzinger P, Greget M, Kessler L, Moulin B. Atypical hemolytic and uremic syndrome due to C3 mutation in pancreatic islet transplantation: a case report. BMC Nephrol. 2020 Sep 19;21(1):405. doi: 10.1186/s12882-020-02062-7. PMID 32950058
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882
- [Derived] Lablanche S, Vantyghem MC, Kessler L, Wojtusciszyn A, Borot S, Thivolet C, Girerd S, Bosco D, Bosson JL, Colin C, Tetaz R, Logerot S, Kerr-Conte J, Renard E, Penfornis A, Morelon E, Buron F, Skaare K, Grguric G, Camillo-Brault C, Egelhofer H, Benomar K, Badet L, Berney T, Pattou F, Benhamou PY; TRIMECO trial investigators. Islet transplantation versus insulin therapy in patients with type 1 diabetes with severe hypoglycaemia or poorly controlled glycaemia after kidney transplantation (TRIMECO): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Jul;6(7):527-537. doi: 10.1016/S2213-8587(18)30078-0. Epub 2018 May 15. PMID 29776895